CLINICAL TRIAL: NCT04843852
Title: Augmentation of Humoral Immunity Using Toll-Like Receptor (TLR) 9 Adjuvanted HBV Surface Antigen to Enhance Anti-HBSAg Response
Brief Title: TLR-9 Adjuvanted Vaccination for Chronic Hepatitis B
Acronym: BOOST-9
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Lydia Tang, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00115083
Record Dates: First submitted 2021-04-06; First posted 2021-04-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hepatitis B; Chronic Hepatitis B
Keywords: hepatitis B; Toll-like receptor; vaccine; hepatitis B surface antibody; HBsAb; anti-HBsAg; hepatitis B surface antigen; HBsAg; TLR9; CpG
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — Hepatitis B Vaccines; Heplisav-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): HEPLISAV-B is available in pre-filled, single-dose 0.5 mL vials. Each dose contains 20 μg of HBsAg and 3,000 μg of 1018 adjuvant. HEPLISAV-B is administered as an intramuscular injection in the deltoid region.
  Study subjects will receive a total of 2 injections, each administered at least 4 weeks apart - the same dosing schedule recommended for hepatitis B prevention.
  Once enrolled, participants will have study visits on days 0 (first injection), and weeks 2, 4 (second injection), 8, and 28. They will also have phone follow ups on day 7 and week 5 (7 days after each injection) and week 56 (end of study).
  Interventions: Drug: Hepatitis B Vaccine Recombinant, Adjuvanted Intramuscular Solution [HEPLISAV-B]

INTERVENTIONS:
Drug: Hepatitis B Vaccine Recombinant, Adjuvanted Intramuscular Solution [HEPLISAV-B] — one 0.5ml intramuscular injection on day 0 and week 4.

SUMMARY:
The goal of this clinical trial is to learn if HEPLISAV-B, a vaccine that is approved to prevent hepatitis B infection in people that are not already infected, is safe in people already chronically infected with hepatitis B. The main quiestions it aims to answer are:

1. Is HEPLISAV-B safe in people with chronic hepatitis B?
2. What side effects, if any, could HEPLISAV-B cause in people with chronic hepatitis B?
3. How does HEPLISAV-B affect the cells that fight chronic hepatitis B?

Participants will:

* Receive HEPLISAV-B as an injection in the muscle, one injection every 4 weeks, for a total of 2 injections.
* Visit the clinic a total of 5 times, and have 3 phone follow ups over 14 months.
* Be asked if they are having any side effects from HEPLISAV-B.
* Have blood samples collected.

DETAILED DESCRIPTION:
Ten people with chronic hepatitis B and virally suppressed on nucleos(t)ide analogue (NUC) therapy will receive a total of two 0.5ml intramuscular injections of HEPLISAV-B, a CpG-adjuvanted vaccine, the first injection on day 0, and the second injection on week 4.

Participants will visit the clinic on day 0, and weeks 2, 4, 8, and 28. They will also have phone follow ups on day 7, and weeks 5 and 56. At each follow up, participants will be asked about any side effects. At each clinic visit blood samples will be collected. For 7 days after each HEPLISAV-B injection, participants will complete a diary to document any reactions to the injection.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, an individual must meet all the following criteria:

1. >18 years old
2. Diagnosed with CHB infection, without HIV, hepatitis C nor hepatitis D co-infections
3. Currently receiving NUC with HBV VL <100 IU/ml for ≥ 12 months
4. Willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, and other study procedures.
5. Determined by medical history, targeted physical examination, and clinical judgement of the investigator to be in good health.

CHB infection is defined as any individual with documentation of a positive HBsAg and/or detectable HBV DNA test for at least 6 months.

Exclusion Criteria:

A participant will be ineligible to participate on this study if any of the following criteria are met:

1. Pregnancy or breast feeding.
2. Received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening (for corticosteroids ≥ 20 mg/day of prednisone equivalent). Received anti-CD20 immunosuppressant within 12 months of screening. Topical tacrolimus is allowed if not used within 14 days prior to Day 1.
3. Received or plans to receive live virus vaccines within 4 weeks, and inactivated vaccine within 2 weeks prior to randomization; or plans to receive a non-study vaccine within 28 days after any dose of study vaccine (with exception for seasonal influenza vaccine within 14 days of study vaccine).
4. Administration of any blood products within 3 months prior to randomization.
5. Participation in a study with an investigational study product or device within 30 days of randomization.
6. Has allergies to any hepatitis B and/or yeast-based vaccines.
7. Subjects meeting any of the following laboratory parameters at screening:

   1. ALT greater than 3 times the upper limit of normal
   2. Elevated total bilirubin WITH direct bilirubin greater than 2 times upper limit of normal
8. Is acutely ill or febrile 72 hours prior to or at vaccine dosing (fever defined as ≥ 38.0°C/100.4°F). Participants meeting this criterion may be rescheduled within the relevant window periods. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator.
9. Have any chronic or acute or unstable conditions that the investigator considers a contraindication to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety and reactogenicity of the Hepatitis B Virus Surface Antigen, Recombinant (HEPLISAV-B; Dynavax Technologies Corporation) Vaccine in patients with chronic hepatitis B | Baseline to 7 days following each vaccine dose
  Number of local and systemic solicited adverse events
Occurence of unsolicited adverse events | from dose 1 to 28 days following each vaccine dose
  Number of unsolicited adverse events
Medically Attended Adverse Events | From first vaccine to 12 months after last vaccine on study.
  Number of Medically Attended Adverse Events (MAAEs)

OTHER OUTCOMES:
Change in hepatitis B surface antigen levels | Day 0 to week 28
  Hepatitis B surface antigen levels (international units per milliliter, IU/mL) will be measured at baseline, and thoughout study
Anti-HBsAg Seroconversion | Day 0 through 12 months post vaccination
  Number of patients with anti-HBsAg seroconversion
Changes in immunologic and virologic responses throughout study | baseline to week 28
  Change in hepatitis B surface antigen-specific immune cell types (percentage of cells) and function (percentage of cells producing cytokines), and hepatitis B virus viral markers (international units per milliliter, IU/mL) will be evaluated at baseline, and throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Tang, MBChB, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Institute of Human Virology, University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No